CLINICAL TRIAL: NCT04507256
Title: A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD7442 in Healthy Adults
Brief Title: AZD7442 - a Potential Combination Therapy for the Prevention and Treatment of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8850C00001; 2020-003076-40 (EudraCT Number)
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Results first posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
Keywords: Coronavirus; Severe acute respiratory syndrome coronavirus 2; Pharmacokinetics; Safety and tolerability
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be blinded for all placebo controlled dose groups, ie, the Principal Investigator (PI), all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD7442 (Experimental): Participants will receive AZD7442 doses across five fixed-dose cohorts via intravenous (IV) infusions (three cohorts will be administered sequentially, and one cohort will receive co-administration of AZD8895 + AZD1061, mixed into a single infusion) and direct gluteal intramuscular (IM) injections (administered sequentially).
  Interventions: Combination Product: AZD7442
- Placebo (Placebo Comparator): Placebo will be administered to participants across five fixed-dose cohorts similar to the active treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: AZD7442 — Participants randomized to AZD7442 will be administered dose 1, each in Cohort 1a (IM) and Cohort 1b (IV). Participants in Cohort 2 and 3 will receive AZD7442 (IV) doses 2 and 3, respectively. Participants in Cohort 4 will receive AZD7442 (IV) dose 4.
  Arms: AZD7442
Other: Placebo — Participants randomised to placebo will receive the same volume of solution as participants on active treatment.
  Arms: Placebo

SUMMARY:
In this first-in-humans dose escalation study, AZD7442 (AZD8895 + AZD1061) will be evaluated for safety, tolerability, pharmacokinetics, and generation of anti-drug antibodies (ADAs). The study is intended to enable future studies of AZD7442's efficacy in preventing and treating COVID-19.

DETAILED DESCRIPTION:
This is a Phase I, first time in human, randomised, double-blind, placebo-controlled, and dose escalation study.

The study will comprise of:

1. A Screening Period of up to 27 days (Day -28 through Day -2);
2. A Treatment Period during which participants will be resident at the Clinical Unit from Day -1, 1 day before Investigational Medicinal Product (IMP) administration (on Day 1) until at least 24 hours after IMP administration, will be discharged on Day 2 after all safety evaluations have been completed, and
3. A Follow up Period lasting 360 days (through to Day 361) after the IMP dose.

The study will be conducted at a single study centre in United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally required authorisation obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.
* Negative SARS-CoV-2 qRT-PCR and/or serology tests prior to randomisation.
* Weight ≥ 50 kg and ≤ 110 kg at screening, including a BMI of ≥ 18.0 to ≤ 30.0 kg/m^2.
* Healthy by medical history, physical examination, and baseline safety laboratory studies, according to the judgement of the PI.
* Electrocardiogram without clinically significant abnormalities at screening.
* Able to complete the Follow-up Period through Day 361.
* Females of childbearing potential who are sexually active with a non-sterilised male partner must have used a highly effective method of contraception for at least 28 days prior to dosing with IMP and must agree to continue using such precautions until the Final Follow-up Visit. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception.

Exclusion Criteria:

* Known hypersensitivity to any component of the IMP.
* History of allergic disease or reactions likely to be exacerbated by any component of the IMP.
* Previous hypersensitivity, infusion-related reaction or severe adverse reaction following administration of a mAbs.
* Acute (time-limited) illness, including fever above 37.5°C (99.5 °F), on day prior to or day of planned dosing; participants excluded for transient acute illness may be dosed if illness resolves within the 27-day Screening Period or may be rescreened once.
* Any drug therapy within 7 days prior to Day 1 (except contraceptives or a single use of acetaminophen, aspirin, antihistamine, or combination over the counter (OTC) product that contains acetaminophen with an antihistamine, or OTC nonsteroidal anti-inflammatory agent at a dose equal to or lower than that recommended on the package). Vitamins and other nutritional supplements that are not newly introduced, ie, have been taken for at least 30 days prior to enrolment, are not exclusionary.
* Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 2 months prior to screening.
* Receipt of immunoglobulin or blood products within 6 months prior to screening.
* SARS CoV-2 or COVID-19:

  * Participants with any confirmed current or previous COVID-19 infection before randomisation.
  * Participant has clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnoea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
  * Any prior receipt of investigational or licensed vaccine indicated for the prevention of SARS CoV-2 or COVID-19 or expected receipt during the period of study follow up.
* Receipt of any IMP in the preceding 90 days or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study.
* Previous receipt of a mAb within 6 months, or five antibody half lives (whichever is longer), prior to study start.
* Immunodeficiency due to illness, including Human immunodeficiency virus (HIV) infection, or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening. HIV testing must be negative at screening.
* Either history of active infection with hepatitis B or C or positive test for hepatitis C or for hepatitis B surface antigen at screening.
* History of infection with SARS or MERS.
* Aspartate aminotransferase, ALT, or serum creatinine above the ULN; bilirubin and ALP >1.5 × ULN.
* Haemoglobin or platelet count below the LLN at screening. White blood cell or neutrophil count outside normal references ranges.
* History of malignancy.
* Any laboratory value in the screening panel that, in the opinion of the PI, is clinically significant or might confound analysis of study results.
* Pregnant or nursing female.
* History of alcohol or drug abuse within the past 2 years that, according to the PI, might affect assessments of safety or ability of participant to comply with all study requirements OR positive urine drug or alcohol screening.
* Any condition that, in the opinion of the PI, might compromise participant safety or interfere with evaluation of the IMP or interpretation of participant safety or study results.
* Employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
* Absence of suitable veins for blood sampling (IM and IV cohorts) and administration of IMP (IV cohorts).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, MD, MSc, PhD, Principal Investigator — Parexel EPCU (London)
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Forte-Soto P, Albayaty M, Brooks D, Arends RH, Tillinghast J, Aksyuk AA, Bouquet J, Chen C, Gebre A, Kubiak RJ, Pilla Reddy V, Seegobin S, Streicher K, Templeton A, Esser MT. Safety, Tolerability and Pharmacokinetics of Half-Life Extended Severe Acute Respiratory Syndrome Coronavirus 2 Neutralizing Monoclonal Antibodies AZD7442 (Tixagevimab-Cilgavimab) in Healthy Adults. J Infect Dis. 2023 May 12;227(10):1153-1163. doi: 10.1093/infdis/jiad014. PMID 36683419
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00001&attachmentIdentifier=fed309b0-1256-498b-9881-da887ad7f778&fileName=__CSR_Full_18_Mar_2022_D8850C00001_(CSR_Synopsis)_Redacted.pdf&versionIdentifier=
- See also: Redacted CSP and SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00001&attachmentIdentifier=c3a63805-65d0-4dfe-a038-d159f873ea1c&fileName=d8850c00001-csp-amendment-6-final_(redacted)_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 healthy participants were enrolled at a single study center in the United Kingdom (UK) from 18 August 2020 to 19 0ctober 2021.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. A washout period was not included in this study.
Groups:
- Pooled Placebo: Participants received single intravenous infusion (IV) or intramuscular injection (IM) of placebo.
- AZD7442 300 mg, IM: Participants received 300 mg of AZD7442 (AZD8895 + AZD1061) via intramuscular injection (IM) administered in 2 sequential injections, starting with 150 mg AZD8895 and followed by 150 mg AZD1061.
- AZD7442 300 mg, IV: Participants received 300 mg of AZD7442 (AZD8895 + AZD1061) via intravenous infusion (IV) administered in 2 sequential infusions, starting with 150 mg AZD8895 and followed by 150 mg AZD1061.
- AZD7442 1000 mg, IV: Participants received 1000 mg of AZD7442 (AZD8895 + AZD1061) via IV infusion administered in 2 sequential infusions, starting with 500 mg AZD8895 and followed by 500 mg AZD1061.
- AZD7442 3000 mg, IV: Participants received 3000 mg of AZD7442 (AZD8895 + AZD1061) via IV infusion administered in 2 sequential infusions, starting with 1500 mg AZD8895 and followed by 1500 mg AZD1061.
- AZD7442 3000 mg, IV Co-administered: Participants received 3000 mg of AZD7442 (AZD8895 + AZD1061) via IV infusion, the investigational medicinal product (IMP) was co-administered as a single IV infusion containing both (1500 mg of AZD8895 and 1500 mg of AZD1061).
Period: Overall Study
Arm/Group | Pooled Placebo | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 10 | 9 | 10 | 10
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set consisted of all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (11.45) | 41.9 (6.51) | 40.7 (7.83) | 38.9 (8.86) | 35.8 (9.44) | 39.6 (9.30) | 39.17 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 6 | 3 | 3 | 4 | 23
  Male | 5 | 8 | 4 | 7 | 7 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 10 | 9 | 10 | 10 | 10 | 10 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 0 | 3 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 0 | 1 | 5
  White | 6 | 6 | 7 | 8 | 6 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: The safety and tolerability of AZD7442 administered IV or IM to healthy adult participants 18 to 55 years of age was evaluated.
Time Frame: From screening day (Day -28) until Follow-up/end of treatment visit (Day 361)
Population: Safety analysis set included all participants who were randomized and received any amount of AZD7442.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants
  Any AE | 8 | 2 | 5 | 6 | 7 | 6
  Any AE with outcome of death | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome of death) | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of Investigational Medicinal Product (IMP) | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to dose interruption | 0 | 0 | 0 | 0 | 1 | 0
  Ant AE leading to dose reduction | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to withdrawal from the study | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Serum Concentration (Cmax) of AZD7442
Description: The single dose Cmax of AZD7442 and of the individual monoclonal antibodies (mAbs) in serum were evaluated.
Time Frame: Day 1 (pre-dose, 8 h), Day 2 (24 h), Day 4 (72 h), Day 6 (120 h), Day 8 (168), Day 15 (336 h), Day 31 (720 h), Day 61 (1440 h), Day 91 (2160 h), Day 151 (3600 h), Day 211 (5040), Day 271 (6480 h), and Day 361 (8640 h)
Population: The Pharmacokinetic (PK) analysis set consisted of all participants in the safety analysis set who received AZD7442 and who had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL (microgram per milliliter)
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 10
μg/mL (microgram per milliliter)
  AZD8895 | 16.52 (35.56) | 53.71 (10.24) | 162.2 (11.31) | 505.8 (10.54) | 447.8 (8.980)
  AZD1061 | 15.27 (38.53) | 51.69 (12.31) | 154.3 (14.66) | 465.5 (11.09) | 419.3 (11.62)

3. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of AZD7442
Description: The single dose tmax of AZD7442 and of the individual mAbs in serum was evaluated
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all participants in the safety analysis set who received AZD7442 and who had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data.
Measure: Median (Full Range); unit: Day
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Day
  AZD8895 | 13.96 [3.05 to 29.99] | 0.04 [0.02 to 0.33] | 0.04 [0.02 to 0.05] | 0.10 [0.06 to 0.13] | 0.05 [0.05 to 0.05]
  AZD1061 | 13.98 [3.05 to 60.23] | 0.02 [0.02 to 0.96] | 0.02 [0.02 to 0.34] | 0.06 [0.06 to 0.33] | 0.05 [0.05 to 0.33]

4. Secondary Outcome: Terminal Elimination Half-life (t½λz) of AZD7442
Description: The single dose t½λz of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10
Day
  AZD8895 | 87.76 (14.56) | 86.97 (5.195) | 92.38 (17.23) | 91.27 (7.827) | 95.33 (11.06)
  AZD1061 | 79.78 (9.649) | 91.08 (9.152) | 83.05 (16.22) | 88.52 (9.086) | 87.17 (10.78)

5. Secondary Outcome: Area Under the Concentration Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of AZD7442
Description: The single dose AUClast of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL (microgram per milliliter)
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10
day*μg/mL (microgram per milliliter)
  AZD8895 | 2367 (28.92) | 3467 (13.20) | 9237 (11.75) | 29800 (9.799) | 29380 (10.81)
  AZD1061 | 2018 (30.98) | 3085 (13.01) | 9245 (11.22) | 28160 (10.85) | 28210 (11.21)

6. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve Extrapolated to Infinity (AUCinf) of AZD7442
Description: The single dose AUCinf of AZD7442 and of the individual mAbs in serum was evaluated. The bioavailability (F) of AZD7442 Dose 1 administered by IM was calculated as the ratio of geometric mean AUCinf after IM to IV, for mAb AZD8895 and mAb AZD1061 is also presented.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL (microgram per milliliter)
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10
day*ug/mL (microgram per milliliter)
  AZD8895 | 2526 (29.75) | 3677 (13.75) | 9893 (12.58) | 31850 (10.85) | 31850 (11.89)
  AZD1061 | 2130 (31.25) | 3276 (14.17) | 9712 (11.69) | 29860 (11.71) | 30030 (11.82)
Statistical Analysis 1: Comparison: AZD7442 300 mg, IM vs AZD7442 300 mg, IV; Bioavailability of AZD8895 at the end of study (Day 361); Test type: Other — Bioavailability; Ratio of geometric mean AUCinf = 68.69 — The bioavailability of AZD7442 Dose 1 administered by IM was, calculated as the ratio of geometric mean AUCinf after IM to IV, for mAb AZD8895
Statistical Analysis 2: Comparison: AZD7442 300 mg, IM vs AZD7442 300 mg, IV; Bioavailability of AZD1061 at the end of study (Day 361); Test type: Other — Bioavailability; Ratio of geometric mean AUCinf = 65.02 — The bioavailability of AZD7442 Dose 1 administered by IM was, calculated as the ratio of geometric mean AUCinf after IM to IV, for mAb AZD1061

7. Secondary Outcome: Systemic Clearance (CL) of AZD7442 IV Infusion
Description: The single dose CL of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all participants in the safety analysis set who received AZD7442 and who had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data. It was pre-specified in the statistical analysis plan (SAP) and clinical study protocol (CSP) to report CL for only arms receiving IV infusion.
Measure: Mean (Standard Deviation); unit: L (Litre)/day
Arm/Group | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 9 | 9 | 10 | 10
L (Litre)/day
  AZD8895 | 0.04113 (0.005411) | 0.05090 (0.006510) | 0.04736 (0.005317) | 0.04740 (0.005661)
  AZD1061 | 0.04618 (0.006162) | 0.05180 (0.006260) | 0.05055 (0.006086) | 0.05026 (0.006036)

8. Secondary Outcome: Apparent Total Clearance (CL/F) of AZD7442 IM Injection
Description: The single dose CL/F of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all participants in the safety analysis set who received AZD7442 and who had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data. It was pre-specified in the SAP and CSP to report CL/F for only arm receiving IM injection.
Measure: Mean (Standard Deviation); unit: L (Litre)/day
Arm/Group | AZD7442 300 mg, IM
Number analyzed (Participants) | 10
L (Litre)/day
  AZD8895 | 0.06174 (0.01857)
  AZD1061 | 0.07383 (0.02733)

9. Secondary Outcome: Apparent Volume of Distribution at Terminal Phase (Vz/F) of AZD7442
Description: The single dose Vz/F of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L (Litre)
Arm/Group | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 9 | 9 | 10 | 10
L (Litre)
  AZD8895 | 7.771 (2.152) | 5.150 (0.5804) | 6.814 (1.065) | 6.227 (0.5926) | 6.514 (0.7232)
  AZD1061 | 8.471 (2.832) | 6.042 (0.5914) | 6.241 (0.9723) | 6.449 (0.6920) | 6.324 (0.7784)

10. Secondary Outcome: Volume of Distribution at Steady State (Vss) of AZD7442 IV Infusion
Description: The single dose Vss of AZD7442 and of the individual mAbs in serum was evaluated.
Time Frame: as for outcome 2
Population: The PK analysis set consisted of all participants in the safety analysis set who received AZD7442 and who had evaluable serum PK data, with no important protocol deviations thought to impact on the analysis of the PK data. It was pre-specified in the SAP and CSP to report Vss for only arms receiving IV infusion.
Measure: Mean (Standard Deviation); unit: L (Litre)
Arm/Group | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 9 | 9 | 10 | 10
L (Litre)
  AZD8895 | 5.074 (0.4766) | 6.520 (0.9739) | 6.118 (0.5983) | 6.373 (0.6854)
  AZD1061 | 5.687 (0.4691) | 6.020 (0.8755) | 6.311 (0.6722) | 6.286 (0.7465)

11. Secondary Outcome: Percentage of Participants Who Have Positive Antidrug Antibodies (ADA) of AZD8895 and AZD1061
Description: The ADA response to AZD7442 in serum was evaluated.
Time Frame: Day 361 (Post dose)
Population: Safety analysis set included all participants who were randomized and received any amount of AZD7442.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
Participants
  AZD8895 | 0 | 1 | 0 | 0 | 0 | 0
  AZD1061 | 0 | 4 | 3 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening day (Day -28) until Follow-up/end of treatment visit (Day 361)
Arm/Group | Pooled Placebo | AZD7442 300 mg, IM | AZD7442 300 mg, IV | AZD7442 1000 mg, IV | AZD7442 3000 mg, IV | AZD7442 3000 mg, IV Co-administered
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 8/10 | 2/10 | 5/10 | 6/10 | 7/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=10) | AZD7442 300 mg, IM (N=10) | AZD7442 300 mg, IV (N=10) | AZD7442 1000 mg, IV (N=10) | AZD7442 3000 mg, IV (N=10) | AZD7442 3000 mg, IV Co-administered (N=10)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myxoid cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT04507256/Prot_SAP_000.pdf